CLINICAL TRIAL: NCT03338426
Title: A Randomized, Double-blind, Multicenter, Phase III Study to Evaluate the Efficacy and Safety of Combination Treatment of Fimasartan/Atorvastatin in Patients With Essential Hypertension and Dyslipidemia
Brief Title: A Study to Evaluate the Efficacy and Safety of Combination Treatment of Fimasartan/Atorvastatin in Patients With Essential Hypertension and Dyslipidemia
Acronym: FIESTA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BR-FAVC-CT-301
Record Dates: First submitted 2017-10-30; First posted 2017-11-09 (Actual); Last update posted 2019-11-05 (Actual); Status verified 2019-10

CONDITIONS: Essential Hypertension, Dyslipidemia
MeSH Terms: conditions — Essential Hypertension; Dyslipidemias | interventions — fimasartan; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental (Experimental): Co-administration of a fixed dose combination of Fimasartan 120mg and Atorvastatin 40mg
  Interventions: Drug: Fimasartan 120mg; Drug: Atorvastatin 40mg
- Active Comparator 1 (Active Comparator): Co-administration of Fimasartan 120mg and Placebo for Atorvastatin 40mg
  Interventions: Drug: Fimasartan 120mg; Drug: Placebo for Atorvastatin 40mg
- Active Comparator 2 (Active Comparator): Co-administration of Atorvastatin 40mg and Placebo for Fimasartan 120mg
  Interventions: Drug: Atorvastatin 40mg; Drug: Placebo for Fimasartan 120mg

INTERVENTIONS:
Drug: Fimasartan 120mg — Fimasartan 120mg will be administrated once daily for 8 weeks treatment period
  Arms: Active Comparator 1; Experimental
Drug: Atorvastatin 40mg — Atorvastatin 40mg will be administrated once daily for 8 weeks treatment period
  Arms: Active Comparator 2; Experimental
Drug: Placebo for Fimasartan 120mg — Placebo for Fimasartan 120mg will be administrated once daily for 8 weeks treatment period
  Arms: Active Comparator 2
Drug: Placebo for Atorvastatin 40mg — Placebo for Atorvastatin 40mg will be administrated once daily for 8 weeks treatment period
  Arms: Active Comparator 1

SUMMARY:
The objective of this clinical study is to evaluate the efficacy and safety by comparing the fimasartan/atorvastatin treatment group to the fimasartan/placebo treatment group and the placebo/atorvastatin treatment group respectively at Week 8 in patients with essential hypertension and dyslipidemia.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily provided a written consent to participate in this clinical study
2. Male or female adults aged 19-70 years
3. Patients must have been confirmed essential hypertension and dyslipidemia at Screening visit (V1)
4. Uncontrolled blood pressure (140 mmHg ≤ mean SiSBP < 180 mmHg) at the pre- baseline visit (V2) after wash-out period
5. Able to understand this study, be cooperative in the execution of the study, and participate in the study until its completion

Exclusion Criteria:

1. Severe hypertension with mean Sitting systolic blood pressure(SiSBP)≥180 mmHg or Sitting diastolic blood pressure(SiDBP) ≥110 mmHg at the screening visit (V1) and the pre-baseline visit (V2), or orthostatic hypotension accompanied by symptoms
2. Difference of Sitting systolic blood pressure(SiSBP) ≥ 20 mmHg and Sitting diastolic blood pressure(SiDBP) ≥ 10 mmHg between Lt and Rt arms for 3 consecutive times at the screening visit (V1)
3. Secondary hypertension patients: Secondary hypertension is not limited to the following diseases; (e.g., renovascular disease, adrenal medullary and cortical hyperfunctions, coarctation of the aorta, hyperaldosteronism, unilateral or bilateral renal artery stenosis, Cushing's syndrome, pheochromocytoma, and polycystic kidney disease)
4. Uncontrolled diabetes mellitus (currently on insulin, or HbA1c >9% at the pre-baseline visit (V2)), or uncontrolled hypothyroidism (TSH ≥1.5 times the upper limit at the pre-baseline visit (V2))
5. Heart disease (heart failure of New York Heart Association (NYHA) class 3 and 4), or ischemic heart disease (angina pectoris, myocardial infarction), peripheral vascular diseasenewly diagnosed within 6 months prior to the screening visit (V1), percutaneous transluminal coronary angioplasty, or coronary artery bypass graft, etc.
6. Clinically significant ventricular tachycardia, atrial fibrillation, atrial flutter; or other arrhythmia conditions that are determined to be clinically significant by the investigator
7. Hypertrophic obstructive cardiomyopathy, severe obstructive coronary artery disease, aortic stenosis, or hemodynamically significant aortic valve stenosis or mitral valve stenosis
8. Cerebrovascular disorder (stroke, cerebral infarction, transient cerebral ischemic attack, cerebral hemorrhage, etc. within 6 months prior to the screening visit (V1)
9. Pregnant or lactating women

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-04-22 (Actual); Study Completion 2019-04-22 (Actual)

PRIMARY OUTCOMES:
SiSBP | 8weeks from Baseline Visit
  The change in Sitting systolic blood pressure(SiSBP) from baseline in the test group(Fimasartan 120mg/Atorvastatin 40mg) at Week 8 compared to the Active Comparator group 2(Atorvastatin 40mg)
LDL-C | 8weeks from Baseline Visit
  The change in LDL-C from baseline in the test group at Week 8 compared to the active comparator group 1(fimasartan 120 mg)

SECONDARY OUTCOMES:
SiSBP | 8weeks from Baseline Visit
  The change in Sitting systolic blood pressure(SiSBP) from baseline in the test group(Fimasartan 120mg/Atorvastatin 40mg) at Week 8 compared to the Active Comparator group 1(Fimasartan 120mg)
LDL-C | 8weeks from Baseline Visit
  The change in LDL-C from baseline in the test group(Fimasartan 120mg/Atorvastatin 40mg) at Week 8 compared to the Active Comparator group 2(Atorvastatin 40mg)

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, South Korea